CLINICAL TRIAL: NCT00004805
Title: Study of the Effect of Four Methods of Cardiopulmonary Resuscitation Instruction on Psychosocial Response of Parents With Infants at Risk of Sudden Death
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, Los Angeles (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Educational/Counseling/Training
Other Study IDs: 199/11973; UCLA-94061792
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-02

CONDITIONS: Pulmonary Hypertension; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome
Keywords: bronchopulmonary dysplasia; cardiovascular and respiratory diseases; disease-related problem/condition; educational needs; hypertensive disorder; neonatal disorders; primary pulmonary hypertension; rare disease; respiratory distress syndrome
MeSH Terms: conditions — Hypertension, Pulmonary; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Respiratory Tract Diseases; Hypertension; Infant, Newborn, Diseases; Familial Primary Pulmonary Hypertension; Rare Diseases

INTERVENTIONS:
Behavioral: CPR instruction

SUMMARY:
OBJECTIVES: I. Describe the psychosocial response of parents and caretakers who learn cardiopulmonary resuscitation (CPR) techniques for infants at high risk for respiratory or cardiac arrest.

II. Compare the effect of 4 methods of CPR instruction on psychosocial response.

III. Evaluate a psychological intervention based on social support theory designed to offset the potential adverse psychological outcomes of CPR instruction.

IV. Evaluate a self-paced CPR learning module using the principles of adult learning theory.

V. Document the level of CPR knowledge and skill retention over time. VI. Document the frequency of CPR and its outcome following a witnessed respiratory or cardiac arrest.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Parents of high-risk infants are randomly assigned to 1 of 4 groups; groups are alternated at each site and the sequence of groups at each site is randomly assigned.

The first group receives a 90-minute, 1-person cardiopulmonary resuscitation (CPR) and obstructed airways management instruction.

The second group receives the same instruction plus a 1-hour social support discussion. Ongoing support is provided with weekly phone calls to assess caretaker status and answer questions regarding the infant's health.

The third group learns CPR using a self-paced multimedia learning module. The control group receives the standard CPR instruction at hospital discharge. Participants are followed at 2 weeks, then at 3 and 6 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Population Characteristics-- Parent or caretaker with infant at risk for sudden death, i.e.: Birth weight less than 2500 g Abnormal pneumogram Bronchopulmonary dysplasia Respiratory distress syndrome Primary pulmonary hypertension Congenital cardiac abnormality Home oxygen requirement Asphyxia or hypoxia Apnea of infancy Documented episode of apnea or bradycardia Sibling of sudden infant death syndrome victim Substance-abusing mother Literate in Spanish or English No history of mental illness No contraindication to cardiopulmonary resuscitation instruction, e.g., arthritis or orthopedic injury No cardiopulmonary resuscitation instruction within 2 years

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 1991-09; Study Completion 1997-08

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Dracup, Study Chair — University of California, Los Angeles